CLINICAL TRIAL: NCT03294174
Title: Opioid Induced Loss of Local Anesthetic Potency in Patients Undergoing Total Knee
Brief Title: Opioid Induced Loss of Local Anesthetic Potency in Patients Undergoing Total Knee Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: Responsible Investigator left institution
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO15020146
Record Dates: First submitted 2016-04-10; First posted 2017-09-26 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2017-10

CONDITIONS: Opioid Tolerance, Opioid Naive, Opioid Exposure
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Synovial tissues will be collected from each study patient

GROUPS / COHORTS (3):
- Opioid naive: Patients who have not been exposed to opioids, but will receive ropivacaine injection
  Interventions: Drug: Ropivacaine injection
- Opioid exposure: Patients who have been exposed to(> 6months), but not currently taking opioids, but will receive ropicacaine injection
  Interventions: Drug: Ropivacaine injection
- opioid tolerance: Patients who have been actively taking opioids with a tolerant dose based on FDA guideline, but will receive ropivacaine injection
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — Ropivacaine administered to provide nerve block
  Other Names: ropivacaine nerve block

SUMMARY:
Peripheral nerve blocks with local anesthetics (LAs) have become an integral part of postoperative pain management particularly for patients undergoing major limb procedures such as such as Total Knee Arthroplasty (TKA). And while postoperative pain management in patients with a history of chronic opioid use may be difficult with systemic opioids because of opioid tolerance, there is anecdotal evidence suggesting that these patients may also be less responsive to LAs. Preliminary data from pre-clinical animal study show that there is a decreased LA potency in blocking sciatic nerve in opioid tolerant rats. And the decrease in LA potency is reversed by the knock-down of the beta4 subunits of Voltage-gated sodium channels along the sciatic nerves, suggesting the opioid induced intrinsic changes in the peripheral nerve as an underlying mechanism for opioid induced loss of LA potency.

Study Goals: To determine the extent to which the changes in beta4 subunits of voltage-gated sodium channels are reflected in surgical patients.

Experimental Design / methodology: This is a prospective, double-blind, active treatment controlled study. TKA Patients who receive nerve blocks will be grouped according to their history of pre-operative opioid use, and then tested for local anesthetic use for nerve block. Synovial tissues will also be collected for the analysis of beta4 subunits.

Subject population: Patients who are scheduled for TKA procedure, and agree to receive peripheral nerve block for postoperative pain control, will be recruited for the study. Patients will participate in one of the three study groups: opioid naive, opioid history and opioid tolerant. 30 patients for each group with a total of 90 patients will be recruited.

This study will not only determine the extent to which the preclinical findings are reflected in clinical patients, but also identify the underlying mechanisms that may suggest strategies for more effective post-operative pain management in the growing population of opioid tolerant patients

DETAILED DESCRIPTION:
3 groups of patients will be included in this prospective study: opioid naïve, those using opioids at the time of surgery (opioid tolerant), and those with a history of opioid use, but who are not currently on opioids (tolerant history). The FDA guidelines will be used to define the opioid tolerant patients as a patient taking, for 1 week or longer, at least 60 mg oral morphine /day; 25 ug transdermal fentanyl/hour; 30 mg oral oxycodone /day; 8 mg oral hydromorphone /day; 25 mg oral oxymorphone/day, or an equianalgesic dose of any other opioid.

Patients will be recruited based on the inclusion and exclusion criteria (see below). Patients eligible for the study will be identified in the population seen by orthopedic surgeons practicing at UPMC Shadyside Hospital and recruited at the pre-surgery clinic by the research coordinator or PI. Study patients will be asked to sign the informed consent form at that time. Pre-operative pain socres, dose and duration of pre-operative opioid consumption will be collected. Knee function (Knee Society score and the functional scores) will be recorded. Data collection will be performed by the research coordinator or PI.

All study patients will receive pre-operative femoral and sciatic nerve block catheters under ultrasound guidance. This is the standard care for postoperative pain control. Once nerve block catheters are placed, research study will be performed to determined the LA potency prior to surgery using the up-down approach, to avoid the confound of post-operative pain. Femoral nerve catheters will be initially dosed with 10 ml, 0.5% ropivacaine. This dose (50 mg) is to produce a complete block in 50% of the patients based on previous studies (7). This is the standard dose of LA provided through femoral nerve catheters.

The following approaches to increase and decrease the dose of ropivacaine are part of research procedures:

After the completion of the initial catheter bolus, sensory and motor blocks will be evaluated every 2 min for the first 10 min after injection, and then every 5 min until 30 min after injection. Sensory block is assessed by evaluating the presence and absence of response to thermal stimulation applied to the central sensory region of the blocked nerve. Thermal stimulation will be delivered with a 5 X 5 mm contact thermode (Medoc, Minneapolis, MN). Two different heat ramps are used to preferentially activate A-delta or C-fiber primary afferents. As previously reported, rises in temperature of < 2 °C/s activates C-fiber afferents, whereas heat ramps > 2 °C/s results in activation of A-delta primary afferents (8). Fast (3.4 °C/s) and slow (1.0 °C/s) heat ramps are used to increase temperatures from a 35 °C holding temperature to a plateau of 50°C. The plateau temperature is maintained for 10 and 5 s for the fast and slow heat ramps, respectively. The sequence of fast and slow heat stimulation is applied with a three-minute interval between trials to avoid sensitization. Nociceptive block will be confirmed with a pin prick test . Motor block is assessed by the MRC (Muscle Function Council) scale (0, no active contraction; 5 the normal power) of quadriceps muscles. Effective blocks are defined as complete loss of a thermal sensation at fast and slow ramp tests with MRC scale =0.

Each patient's response to the block determine the LA doses for the subsequent patient. Each time, the delivered LA volumes will remain at 10 ml. The doses to be tested on subsequent patients include 100mg, 75 mg, 25 mg and 10 mg ropivacaine. For example, when effective block is achieved within 30 min after the initial injection of 10 ml, 50 mg ropivacaine, the next patient will receive 25 mg ropivacaine. Conversely, when effective block is not observed, the next patient will receive 75 mg of ropivacaine. After the tests, necessary additional LA will be given to the patients to achieve the final LA dose of 100 mg, which should produce complete block in 99% of the patients (ED99). Response probability is estimated for each LA dose and fit to a probit model function. The resulting probability function yields continuous estimates of the response probabilities over the full dose range. From this curve, it is possible to determine the ropivacaine doses needed to produce a complete block in 50% (ED50), 95%(ED95) and 99%(ED99) of the subjects. The nerve block procedures and the data collection will be performed by the fellows of AIPPS (Acute Interventional Perioperative Pain Service), who are blind to the which group the study patients belong to. The study will be performed at the SDS (Same Day Surgery), Shadyside hospital. It will take 30-45 min to complete the study, which allows ample time for surgery preparations.

After completion of the study, patients will receive standard intra- and post-operative care. Intra-operative pain management will consist of acetaminophen (i.v. 1000 mg), fentanyl boluses (total <500 mcg) and/or dilaudid boluses (total < 5 mg). Post-operative pain management will be supplemented with acetaminophen (1000mg, q6h), and oxycodone (5/10 mg, q4h, p.r.n). Nerve block catheter infusions and boluses (bupivacaine 0.0625% 5 ml/h for femoral block, and bupivacaine 0.03%, 3 ml/h for sciatic block) will start in PACU by nursing staff, who are blind to the study. VAS pain scores and motor function assessment will be recorded every hour in the PACU, and every four hours in the in-patient floor by the research coordinator or PI. Postoperative pain will be managed by the AIPPS team, who is blind to the study. Both femoral and sciatic nerve block infusions will be stopped on post-operative day 3.

Synovial tissue will be collected intraoperatively by research coordinator for analysis of the Na+ channel subunit expression. The synovial tissue, which would be discarded as medical waste, will be transferred to BST(Biomedical Science Tower)w1405 (Dr. Michael S. Gold's lab) for analysis. The lab technician, who will be performing the analysis, is blind to the study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Classification 1,2 and 3;
* Age between 18-80;
* Both males and females of all races
* Receive total knee arthroplasty (TKA)
* Agree to receive peripheral nerve blocks for postoperative pain control

Participants of the study will belong to one of the three groups: opioid naive, opioid history (those with a history of opioid use, but who are not currently on opioids) and opioid tolerant (those using opioids at the time of surgery)

Exclusion Criteria:

* Intolerance and/or known allergy to opioids and/or LAs;
* TKA due to trauma;
* Use of general anesthesia for the operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the study will belong to one of the three groups: opioid naive, opioid history (those with a history of opioid use, but who are not currently on opioids) and opioid tolerant (those using opioids at the time of surgery)
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Sensory and motor function loss after nerve block procedures | within first 30 min
  Sensory block is assessed by evaluating the presence and absence of response to thermal stimulation applied to the central sensory region of the blocked nerve, using Medoc 5x5 thermode (see details in description)

SECONDARY OUTCOMES:
pain | within 1 hour
  VAS pain score will be used to assess pain level
sodium channel subunit changes in synovial tissues | Synovial tissues will be extracted within 1 hour after nerve block. Western blotting techniques will be used to quantify the changes in sodium channel subunit level
  changes in sodium channel subunit level

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw data available upon request